CLINICAL TRIAL: NCT03997760
Title: A Phase 1 Randomized, Double-blind, Placebo-controlled, Multicenter, Ascending Dose, Safety and PK/PD Study of SHP655 (rADAMTS13) in Sickle Cell Disease at Baseline Health
Brief Title: A Study of SHP655 (rADAMTS13) in Sickle Cell Disease
Acronym: RAISE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHP655-101
Record Dates: First submitted 2019-06-14; First posted 2019-06-25 (Actual); Results first posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — ADAMTS13 protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TAK-755 (Experimental): Participants with SCD at their baseline health will receive a single intravenous (IV) infusion at one of the 3 dose levels of 40, 80 and 160 International units per kilogram (IU/kg) in a dose escalation manner.
  Interventions: Drug: TAK-755
- Placebo (Placebo Comparator): Participants with SCD at their baseline health will receive placebo matched to TAK-755 of the 3 dose levels of 40 IU/kg, 80 IU/kg, and 160 IU/kg as single IV infusion.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: TAK-755 — Participants will receive TAK-755 as a single IV infusion at one of the 3 dose levels of 40 IU/kg, 80 IU/kg, or 160 IU/kg.
  Other Names: recombinant ADAMTS13; BAX 930; SHP655
  Arms: TAK-755
Other: Placebo — Participants will receive placebo matched to TAK-755 of the 3 dose levels of 40 IU/kg, 80 IU/kg, and 160 IU/kg as single IV infusion.
  Arms: Placebo

SUMMARY:
TAK-755 (previously known as SHP655) is a medicine used to treat sickle cell disease (SCD). The main aim of the study is to measure the safety and tolerability of TAK-755 in SCD participants.

Study participants will receive TAK-755 or placebo on Day 1. Their SCD will be treated by their doctor according to their doctor's usual clinical practice.

During the study, participants will be asked to follow-up on 13 days following SHP655 or placebo administration for safety assessment. Maximum duration of participation is expected to be about 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years at the time of signing the informed consent.
* An understanding, ability, and willingness to fully comply with study procedures and requirements.
* Ability to voluntarily provide written, signed, and dated (personally or via a legally authorized representative) informed consent to participate in the study.
* Male or female with a documented history of HbSS or HbSβo thalassemia (based on clinical record of genetic, electrophoresis, or high-performance liquid chromatography testing).
* Participant currently taking hydroxyurea must be on a stable dosing for 3 months at screening.

Exclusion Criteria:

* The participant was diagnosed with acute VOC in the 21 days before dosing on Day 1.
* The participant has undergone blood transfusion within the last 30 days or blood transfusion on greater than or equal to (>=) 2 occasions in the last 90 days, at Screening Visit.
* The participant has a history of acquired or congenital thrombotic thrombocytopenic purpura.
* The participant has serum creatinine level greater than (>) 1.2 milligrams per deciliter (mg/dL).
* The participant has alanine transaminase >3* upper limit of normal (based on clinical laboratory normal range), direct bilirubin level >2 mg/dL, or indirect bilirubin level >5 mg/dL at the Screening Visit.
* The participant has a hemoglobin level <5 grams per deciliter (g/dL) at the Screening Visit.
* The participant has a platelet count of <100 000/cubic millimeter (mm^3) at the Screening Visit.
* Signs or symptoms of infection requiring treatment with IV antibiotics during the Screening Period.
* The participant has fever with body temperature of >=38.5 degree Celsius (ºC) (101.3 degree Fahrenheit [ºF]) at the Screening Visit or before dosing on Day 1.
* The participant has Acute Chest Syndrome (ACS), diagnosed or strongly suspected, as evidenced by a new infiltrate on chest radiograph, and one or more of the following criteria:

  1. Fever with body temperature >39°C (102.2°F)
  2. Hypoxia (confirmed by arterial blood gases with partial pressure of arterial oxygen (PaO2) <70 millimeter of mercury [mmHg])
  3. Chest pain
  4. Suspicious findings on physical examination (tachypnea, intercostal retraction, wheezing, and/or rales)
* The participant has recently (within the past 28 days, from Screening Visit) undergone major surgery, requires hospitalization, documented serious bacterial infection requiring antibiotic treatment, or significant bleeding.
* The participant has had a recent (within the past 90 days, from Screening Visit) episode of stroke, transient ischemic attack, symptomatic pulmonary hypertension, or seizure.
* Any history of hemorrhagic stroke or bleeding diathesis.
* The participant has received any of the following protocol-restricted medicines: a) systemic steroid therapy within 48 hours before dosing, or there is the expectation that such therapy may be given during the study (inhaled or topical steroids are allowed); b) Anticoagulant or antiplatelet therapy within the past 3 weeks before dosing; c) crizanlizumab within the past 30 days before dosing; d) voxelotor within the past 14 days before dosing.
* For participants receiving chronic or long-acting opioids, a change in dose or pain requiring medical attention in the past 14 days before dosing.
* The participant has a medical or psychiatric condition that, in the opinion of the investigator, may pose a risk to the participant for participation or interfere with the conduct or results of the study.
* The participant has received or plans to receive any other investigational agent within the 4 weeks prior to the study screening visit or during the course of the study.
* There is the expectation that the participant will not be able to be followed for the duration of the study.
* The participant is pregnant or lactating or a female of childbearing potential or male unable or unwilling to comply with birth control methods or abstinence until the end of study visit.
* The participant with active use of illicit drugs (excluding marijuana) and/or alcohol dependence, as determined by the investigator.
* The participant has been administered SHP655 previously.
* Known life-threatening hypersensitivity reaction, including anaphylaxis, to the parent molecule ADAMTS-13, hamster protein, or other constituents of SHP655.
* The participant has a positive test result for hepatitis B surface antigen, or hepatitis C antibody, or human immunodeficiency virus (HIV) antigen/antibody, at the Screening Visit. However, a participant with a hepatitis C antibody and a negative hepatitis C virus ribonucleic acid (RNA) polymerase chain reaction test is not excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (14):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Colorado Sickle Cell Treatment and Research Center, Aurora, Colorado
  - Sickle Cell Center, Denver, Colorado
  - University of Illinois, Chicago, Illinois
  - Ochsner Health System, New Orleans, Louisiana
  - Johns Hopkins University School Of Medicine, Baltimore, Maryland
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - University of Tennessee -- Memphis, Memphis, Tennessee
  - VCU Health - Research Parent, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fe84db2bf003ab47ae1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 9 active sites in the United States from 21 October 2019 to 26 October 2022.
Pre-assignment Details: A total of 19 participants were enrolled and treated in this study.
Groups:
- Placebo: Participants with Sickle Cell Disease (SCD) at their baseline health received a single intravenous (IV) infusion of placebo matched to TAK-755 at 3 dose levels of 40 International units per kilogram (IU/kg), 80 IU/kg, and 160 IU/kg on Day 1 and followed for up to 28 days.
- TAK-755: 40 IU/kg: Participants with SCD at their baseline health received a single IV infusion of TAK-755 at a dose level of 40 IU/kg on Day 1 and followed for up to 28 days.
- TAK-755: 80 IU/kg: Participants with SCD at their baseline health received a single IV infusion of TAK-755 at a dose level of 80 IU/kg on Day 1 and followed for up to 28 days.
- TAK-755: 160 IU/kg: Participants with SCD at their baseline health received a single IV infusion of TAK-755 at a dose level of 160 IU/kg on Day 1 and followed for up to 28 days.
Period: Overall Study
Arm/Group | Placebo | TAK-755: 40 IU/kg | TAK-755: 80 IU/kg | TAK-755: 160 IU/kg
Started | 5 | 4 | 6 | 4
Completed | 5 | 3 | 6 | 4
Not Completed | 0 | 1 | 0 | 0
Not completed — Protocol Deviation | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set (SAS) included all participants randomized and who received any dose of the investigational product (IP).
Groups:
- Placebo: Participants with SCD at their baseline health received a single IV infusion of placebo matched to TAK-755 at 3 dose levels of 40 IU/kg, 80 IU/kg, and 160 IU/kg on Day 1 and followed for up to 28 days.
- Total: Total of all reporting groups
Arm/Group | Placebo | TAK-755: 40 IU/kg | TAK-755: 80 IU/kg | TAK-755: 160 IU/kg | Total
Number analyzed (Participants) | 5 | 4 | 6 | 4 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 6 | 4 | 19
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 3 | 1 | 8
  Male | 2 | 3 | 3 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 4 | 6 | 4 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 4 | 6 | 4 | 19
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this investigational product (IP) or medicinal product. TEAEs were defined as AEs that started or worsened in severity on or after the infusion of IP. A serious TEAEs was any untoward clinical manifestation of signs, symptoms or outcomes (whether considered related to investigational product or not and at any dose) which resulted in death, was life-threatening, required inpatient hospitalization, prolongation of hospitalization, was an important medical event. TEAEs included both serious and non-serious AEs.
Time Frame: From date of signing informed consent up to end of study visit (Day 28)
Population: SAS included all participants randomized and who received any dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TAK-755: 40 IU/kg | TAK-755: 80 IU/kg | TAK-755: 160 IU/kg
Number analyzed (Participants) | 5 | 4 | 6 | 4
Participants
  Participants with TEAEs | 2 | 2 | 4 | 2
  Participants with Serious TEAEs | 0 | 1 | 0 | 0

2. Primary Outcome: Number of Participants Who Developed Positive Binding Anti-ADAMTS13 and Inhibitory Anti-ADAMTS13 Antibodies to TAK-755
Description: Measurement of Anti-ADAMTS13 antibodies can be used to assess whether the body's immune system has been stimulated to react to TAK-755. Binding Anti-ADAMTS13 antibodies measure antibodies that are able to bind to ADAMTS13, whether or not the antibodies have an effect on how well ADAMTS13 works. An inhibitory Anti-ADAMTS13 antibody is antibody that both binds to ADAMTS13 and able to affect how well ADAMTS13 works. Binding and Inhibitory anti-ADAMTS13 antibodies were categorized as pre-existing, treatment-induced, and treatment-boosted. Pre-existing: anti-ADAMTS13 antibodies were detected in the baseline sample prior to infusion with TAK-755. Treatment-induced: no anti-ADAMTS13 antibodies were detected in baseline sample but were detected in any sample drawn after TAK-755 infusion. Treatment-boosted: anti-ADAMTS13 antibodies were pre-existing and were detected at any time after TAK-755 infusion at titers that were at least 4 steps higher than the titers detected before TAK-755 infusion.
Time Frame: From date of signing informed consent up to end of study visit (Day 28)
Population: The SAS included all participants randomized and who received any dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TAK-755: 40 IU/kg | TAK-755: 80 IU/kg | TAK-755: 160 IU/kg
Number analyzed (Participants) | 5 | 4 | 6 | 4
Participants
  Pre-Existing Inhibitory Anti-ADAMTS13 Antibodies | 0 | 0 | 0 | 0
  Treatment-Induced Inhibitory Anti-ADAMTS13 Antibodies | 0 | 0 | 0 | 0
  Treatment-Boosted Inhibitory Anti-ADAMTS13 Antibodies | 0 | 0 | 0 | 0
  Pre-Existing Binding Anti-ADAMTS13 Antibodies | 1 | 1 | 2 | 2
  Treatment-Induced Binding Anti-ADAMTS13 Antibodies | 1 | 1 | 1 | 0
  Treatment-Boosted Binding Anti-ADAMTS13 Antibodies | 0 | 0 | 0 | 0

3. Secondary Outcome: Incremental Recovery (IR) for ADAMTS13 Activity and ADAMTS13 Antigen of TAK-755
Description: IR was defined as the ratio of maximum increase in plasma ADAMTS13 antigen or activity level to TAK-755 dose per body weight. Baseline was defined as the last non-missing measurement obtained prior to the date and time of the first dose of TAK-755. Baseline-adjusted values were used for this analysis. Baseline-adjusted values at each timepoint were calculated as the measured value minus the pre-infusion (baseline) value and results were summarized overall. Here "IU/mL/IU/kg" refers to "International units per milliliter per international units per kilogram".
Time Frame: Baseline (Pre-dose), 0.25, 1, 3, 8, 24, 72, 120, 168, 216, 288, and 648 hours post-dose
Population: The Pharmacokinetic (PK) Analysis Set included all participants who received at least 1 complete dose of TAK-755 or placebo and provided at least 1 concentration measured at a scheduled time post start of infusion for at least 1 of the PK analytes and had no major protocol deviations or events that may affect the integrity of the PK data. Data was not analyzed for PK parameters in the placebo arm where participants did not receive TAK-755.
Measure: Mean (Standard Deviation); unit: IU/mL/IU/kg
Arm/Group | TAK-755: 40 IU/kg | TAK-755: 80 IU/kg | TAK-755: 160 IU/kg
Number analyzed (Participants) | 4 | 5 | 4
IU/mL/IU/kg
  Baseline-adjusted ADAMTS13 Activity | 0.022440 (32.3) | 0.025227 (33.4) | 0.018423 (33.6)
  Baseline-adjusted ADAMTS13 Antigen | 0.021809 (25.8) | 0.021925 (30.1) | 0.022012 (22.2)

4. Secondary Outcome: Observed Maximum Concentration (Cmax) for ADAMTS13 Activity and ADAMTS13 Antigen of TAK-755
Description: Cmax was a measure of the maximum amount of drug in the plasma after the dose was given. Baseline was defined as the last non-missing measurement obtained prior to the date and time of the first dose of TAK-755. Baseline-adjusted values were used for this analysis. Baseline-adjusted values at each timepoint were calculated as the measured value minus the pre-infusion (baseline) value and results were summarized overall.
Time Frame: Baseline (Pre-dose), 0.25, 1, 3, 8, 24, 72, 120, 168, 216, 288, and 648 hours post-dose
Population: The PK Analysis Set included all participants who received at least 1 complete dose of TAK-755 or placebo and provided at least 1 concentration measured at a scheduled time post start of infusion for at least 1 of the PK analytes and had no major protocol deviations or events that may affect the integrity of the PK data. Data was not analyzed for PK parameters in the placebo arm where participants did not receive TAK-755.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: international units per milliliter
Arm/Group | TAK-755: 40 IU/kg | TAK-755: 80 IU/kg | TAK-755: 160 IU/kg
Number analyzed (Participants) | 4 | 5 | 4
international units per milliliter
  Baseline-adjusted ADAMTS13 Activity | 0.90202 (33.5) | 2.0080 (33.2) | 2.9539 (33.6)
  Baseline-adjusted ADAMTS13 Antigen | 0.49848 (27.9) | 1.0382 (30.3) | 2.0392 (22.2)

5. Secondary Outcome: Time to Reach Cmax (Tmax) for ADAMTS13 Activity and ADAMTS13 Antigen of TAK-755
Description: Tmax was a measure of the time to reach the maximum concentration in the plasma after the drug dose. Baseline was defined as the last non-missing measurement obtained prior to the date and time of the first dose of TAK-755. Baseline-adjusted values were used for this analysis. Baseline-adjusted values at each timepoint were calculated as the measured value minus the pre-infusion (baseline) value and results were summarized overall.
Time Frame: Baseline (Pre-dose), 0.25, 1, 3, 8, 24, 72, 120, 168, 216, 288, and 648 hours post-dose
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | TAK-755: 40 IU/kg | TAK-755: 80 IU/kg | TAK-755: 160 IU/kg
Number analyzed (Participants) | 4 | 5 | 4
hour
  Baseline-adjusted ADAMTS13 Activity | 2.16 [0.32 to 3.03] | 1.08 [0.25 to 74.45] | 0.45 [0.32 to 1.18]
  Baseline-adjusted ADAMTS13 Antigen | 0.45 [0.25 to 24.17] | 1.10 [0.28 to 3.48] | 0.83 [0.32 to 1.50]

6. Secondary Outcome: Terminal Half-Life (t1/2) for ADAMTS13 Activity and ADAMTS13 Antigen of TAK-755
Description: t1/2 was the time required for a given drug concentration in the plasma to decrease by 50%. Baseline was defined as the last non-missing measurement obtained prior to the date and time of the first dose of TAK-755. Baseline-adjusted values were used for this analysis. Baseline-adjusted values at each timepoint were calculated as the measured value minus the pre-infusion (baseline) value and results were summarized overall.
Time Frame: Baseline (Pre-dose), 0.25, 1, 3, 8, 24, 72, 120, 168, 216, 288, and 648 hours post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | TAK-755: 40 IU/kg | TAK-755: 80 IU/kg | TAK-755: 160 IU/kg
Number analyzed (Participants) | 4 | 5 | 4
hour
  Baseline-adjusted ADAMTS13 Activity | NA (NA) — Mean and SD were not determined because insufficient number of participants had appropriate number of positive baseline-adjusted concentration data points to determine this PK parameter. | 54.56 (28.230) | 42.22 (9.7253)
  Baseline-adjusted ADAMTS13 Antigen | NA (NA) — Mean and SD were not determined because insufficient number of participants had appropriate number of positive baseline-adjusted concentration data points to determine this PK parameter. | 65.17 (41.728) | 46.88 (16.821)

7. Secondary Outcome: Mean Residence Time From Zero to Infinite (MRT0-Inf) for ADAMTS13 Activity and ADAMTS13 Antigen of TAK-755
Description: The MRT is the average time that the study product stays in the body (or plasma). The MRT0-Inf is defined as the average time from zero (pre-dose) extrapolated to infinite time (MRT0-inf). Baseline was defined as the last non-missing measurement obtained prior to the date and time of the first dose of TAK-755. Baseline-adjusted values were used for this analysis. Baseline-adjusted values at each timepoint were calculated as the measured value minus the pre-infusion (baseline) value and results were summarized overall.
Time Frame: Baseline (Pre-dose), 0.25, 1, 3, 8, 24, 72, 120, 168, 216, 288, and 648 hours post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | TAK-755: 40 IU/kg | TAK-755: 80 IU/kg | TAK-755: 160 IU/kg
Number analyzed (Participants) | 4 | 5 | 4
hour
  Baseline-adjusted ADAMTS13 Activity | NA (NA) — Mean and SD were not determined because insufficient number of participants had appropriate number of positive baseline-adjusted concentration data points to determine this PK parameter. | 118.6 (46.170) | 87.54 (37.734)
  Baseline-adjusted ADAMTS13 Antigen | NA (NA) — Mean and SD were not determined because insufficient number of participants had appropriate number of positive baseline-adjusted concentration data points to determine this PK parameter. | 116.3 (57.699) | 69.48 (23.555)

8. Secondary Outcome: Mean Residence Time From Zero to 72 Hours Post-dose (MRT0-72) of ADAMTS13 Activity and ADAMTS13 Antigen of TAK-755
Description: The MRT is the average time that the study product stays in the body (or plasma) and The MRT0-72 is defined as the average time from zero (predose) to 72 hours post-dose (MRT0-72). Baseline was defined as the last non-missing measurement obtained prior to the date and time of the first dose of TAK-755.
Time Frame: Baseline (Pre-dose), 0.25, 1, 3, 8, 24, and 72 hours post-dose
Population: Since MRT0-72 was considered irrelevant to the objective of the PK, therefore data for this outcome measure was not collected and reported.
Arm/Group | TAK-755: 40 IU/kg | TAK-755: 80 IU/kg | TAK-755: 160 IU/kg
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Area Under the Curve From Zero to Time of Last Quantifiable Concentration (AUC0-Last) for ADAMTS13 Activity and ADAMTS13 Antigen of TAK-755
Description: AUC0-Last was an area under the concentration-time curve from zero (pre-dose) to time of last quantifiable concentration. Baseline was defined as the last non-missing measurement obtained prior to the date and time of the first dose of TAK-755. Baseline-adjusted values were used for this analysis. Baseline-adjusted values at each timepoint were calculated as the measured value minus the pre-infusion (baseline) value and results were summarized overall.
Time Frame: Baseline (Pre-dose), 0.25, 1, 3, 8, 24, 72, 120, 168, 216, 288, and 648 hours post-dose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour* International unit per milliliter
Arm/Group | TAK-755: 40 IU/kg | TAK-755: 80 IU/kg | TAK-755: 160 IU/kg
Number analyzed (Participants) | 4 | 5 | 4
hour* International unit per milliliter
  Baseline-adjusted ADAMTS13 Activity | NA (NA) — Geometric Mean and %CV were not determined because insufficient number of participants had appropriate number of positive baseline-adjusted concentration data points to determine this PK parameter. | 161.5 (28.1) | 137.2 (36.1)
  Baseline-adjusted ADAMTS13 Antigen | 25.96 (32.9) | 79.05 (22.0) | 105.7 (27.7)

10. Secondary Outcome: Area Under the Curve Time Curve From Zero to 72 Hours Post-dose (AUC0-72) for ADAMTS13 Activity and ADAMTS13 Antigen of TAK-755
Description: AUC0-72 was an area under the concentration-time curve from zero (predose) to 72 hours post-dose (AUC0-72). Baseline was defined as the last non-missing measurement obtained prior to the date and time of the first dose of TAK-755. Baseline-adjusted values were used for this analysis. Baseline-adjusted values at each timepoint were calculated as the measured value minus the pre-infusion (baseline) value and results were summarized overall.
Time Frame: Baseline (Pre-dose), 0.25, 1, 3, 8, 24, and 72 hours post-dose
Population: The PK Analysis Set included all participants who received at least 1 complete dose of TAK-775 or placebo and provided at least 1 concentration measured at a scheduled time post start of infusion for at least 1 of the PK analytes and had no major protocol deviations or events that may affect the integrity of the PK data. Data was not analyzed for PK parameters in the placebo arm where participants did not receive TAK-755.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour* International unit per milliliter
Arm/Group | TAK-755: 40 IU/kg | TAK-755: 80 IU/kg | TAK-755: 160 IU/kg
Number analyzed (Participants) | 4 | 5 | 4
hour* International unit per milliliter
  Baseline-adjusted ADAMTS13 Activity | 19.77 (122.3) | 78.44 (36.8) | 92.41 (27.1)
  Baseline-adjusted ADAMTS13 Antigen | 17.91 (22.7) | 42.86 (9.5) | 73.20 (22.0)

11. Secondary Outcome: Area Under the Curve From Zero to Infinite Time (AUC0-Inf) for ADAMTS13 Activity and ADAMTS13 Antigen of TAK-755
Description: AUC0-inf was area under the concentration-time curve from zero (pre-dose) extrapolated to infinite time. Baseline was defined as the last non-missing measurement obtained prior to the date and time of the first dose of TAK-755. Baseline-adjusted values were used for this analysis. Baseline-adjusted values at each timepoint were calculated as the measured value minus the pre-infusion (baseline) value and results were summarized overall.
Time Frame: Baseline (Pre-dose), 0.25, 1, 3, 8, 24, 72, 120, 168, 216, 288, and 648 hours post-dose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour* International unit per milliliter
Arm/Group | TAK-755: 40 IU/kg | TAK-755: 80 IU/kg | TAK-755: 160 IU/kg
Number analyzed (Participants) | 4 | 5 | 4
hour* International unit per milliliter
  Baseline-adjusted ADAMTS13 Activity | NA (NA) — Geometric Mean and %CV were not determined because insufficient number of participants had appropriate number of positive baseline-adjusted concentration data points to determine this PK parameter. | 190.1 (45.3) | 152.5 (46.6)
  Baseline-adjusted ADAMTS13 Antigen | NA (NA) — Geometric Mean and %CV were not determined because insufficient number of participants had appropriate number of positive baseline-adjusted concentration data points to determine this PK parameter. | 88.34 (34.6) | 114.0 (27.5)

12. Secondary Outcome: Systemic Clearance (CL) for ADAMTS13 Activity and ADAMTS13 Antigen of TAK-755
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body. The total systemic clearance after intravenous dose was estimated by dividing the total administered dose by the plasma Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]). Baseline was defined as the last non-missing measurement obtained prior to the date and time of the first dose of TAK-755. Baseline-adjusted values were used for this analysis. Baseline-adjusted values at each timepoint were calculated as the measured value minus the pre-infusion (baseline) value and results were summarized overall.
Time Frame: Baseline (Pre-dose), 0.25, 1, 3, 8, 24, 72, 120, 168, 216, 288, and 648 hours post-dose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour (L/h)
Arm/Group | TAK-755: 40 IU/kg | TAK-755: 80 IU/kg | TAK-755: 160 IU/kg
Number analyzed (Participants) | 4 | 5 | 4
liters per hour (L/h)
  Baseline-adjusted ADAMTS13 Activity | NA (NA) — Geometric Mean and %CV were not determined because insufficient number of participants had appropriate number of positive baseline-adjusted concentration data points to determine this PK parameter. | 37.22 (64.3) | 74.35 (46.8)
  Baseline-adjusted ADAMTS13 Antigen | NA (NA) — Geometric Mean and %CV were not determined because insufficient number of participants had appropriate number of positive baseline-adjusted concentration data points to determine this PK parameter. | 51.28 (66.1) | 54.47 (54.47)

13. Secondary Outcome: Volume of Distribution at Steady State (Vss) for ADAMTS13 Activity and ADAMTS13 Antigen of TAK-755
Description: Vss is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state which is estimated by MRT(0-inf)*CL. Baseline was defined as the last non-missing measurement obtained prior to the date and time of the first dose of TAK-755. Baseline-adjusted values were used for this analysis. Baseline-adjusted values at each timepoint were calculated as the measured value minus the pre-infusion (baseline) value and results were summarized overall.
Time Frame: Baseline (Pre-dose), 0.25, 1, 3, 8, 24, 72, 120, 168, 216, 288, and 648 hours post-dose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | TAK-755: 40 IU/kg | TAK-755: 80 IU/kg | TAK-755: 160 IU/kg
Number analyzed (Participants) | 4 | 5 | 4
liters
  Baseline-adjusted ADAMTS13 Activity | NA (NA) — Geometric Mean and %CV were not determined because insufficient number of participants had appropriate number of positive baseline-adjusted concentration data points to determine this PK parameter. | 3993 (48.2) | 5771 (17.2)
  Baseline-adjusted ADAMTS13 Antigen | NA (NA) — Geometric Mean and %CV were not determined because insufficient number of participants had appropriate number of positive baseline-adjusted concentration data points to determine this PK parameter. | 4682 (8.4) | 3661 (21.7)

14. Secondary Outcome: Change From Baseline in Von Willebrand Factor: Antigen (VWF:Ag) at Specified Timepoints
Description: Von Willebrand factor (vWF or VWF) is a protein that is one of several components of the coagulation system that work together to stop bleeding within the body. VWF:Ag measures the level of von Willebrand factor protein in the blood. The change from baseline in VWF:Ag concentration was measured at different time points. Baseline was defined as the last non-missing measurement obtained prior to the date and time of the dose of IP. Change from baseline was calculated by subtracting the baseline value from the post-dose value.
Time Frame: Baseline (Pre-dose), 0.25, 1, 3, 8, 24, 72, 120, 168, 216, 288, and 648 hours post-dose
Population: Pharmacodynamic analysis set: All participants who received at least 1 complete dose of TAK-755 or placebo and provided at least 1 valid data point post-dose of the respective infusion for at least 1 PD measurement for any of the PD outcome and had no major protocol deviations or events that may have affected the integrity of the PD data. Overall Number of Participants Analyzed refers participants evaluable for this outcome and "number analyzed" refers participants at the specified timepoints.
Measure: Mean (Standard Deviation); unit: Percentage of vWF Ag
Arm/Group | Placebo | TAK-755: 40 IU/kg | TAK-755: 80 IU/kg | TAK-755: 160 IU/kg
Number analyzed (Participants) | 4 | 3 | 6 | 4
Percentage of vWF Ag
  Change at 0.25 hours: number analyzed (Participants) | 4 | 3 | 5 | 3
  Change at 0.25 hours | 5.20 (23.774) | -29.47 (17.719) | -0.96 (32.870) | -16.27 (9.341)
  Change at 1 hour: number analyzed (Participants) | 4 | 3 | 6 | 3
  Change at 1 hour | -9.90 (27.518) | -19.47 (10.161) | 9.50 (20.168) | 4.00 (12.139)
  Change at 3 hours: number analyzed (Participants) | 4 | 3 | 5 | 2
  Change at 3 hours | -7.80 (12.301) | -18.27 (4.670) | -0.30 (22.744) | NA (NA) — Mean and SD were not determined because insufficient number of participants (<=2 participants) had data and therefore, summary statistics could not be performed, as was pre-specified in the analysis plan.
  Change at 8 hours: number analyzed (Participants) | 4 | 3 | 5 | 2
  Change at 8 hours | -8.20 (14.245) | 13.07 (20.433) | -0.24 (15.028) | NA (NA) — Mean and SD were not determined because insufficient number of participants (<=2 participants) had data and therefore, summary statistics could not be performed, as was pre-specified in the analysis plan.
  Change at 24 hours: number analyzed (Participants) | 4 | 3 | 6 | 3
  Change at 24 hours | 0.10 (17.116) | 16.00 (34.113) | 20.42 (18.756) | 2.93 (24.981)
  Change at 72 hours: number analyzed (Participants) | 4 | 3 | 6 | 3
  Change at 72 hours | -25.20 (27.695) | 8.93 (43.275) | 20.32 (25.345) | 9.47 (25.026)
  Change at 120 hours: number analyzed (Participants) | 3 | 2 | 6 | 3
  Change at 120 hours | -14.40 (37.183) | NA (NA) — Mean and SD were not determined because insufficient number of participants (<=2 participants) had data and therefore, summary statistics could not be performed, as was pre-specified in the analysis plan. | 0.67 (29.733) | 9.60 (47.411)
  Change at 168 hours: number analyzed (Participants) | 3 | 2 | 6 | 3
  Change at 168 hours | -46.80 (23.708) | NA (NA) — Mean and SD were not determined because insufficient number of participants (<=2 participants) had data and therefore, summary statistics could not be performed, as was pre-specified in the analysis plan. | 6.82 (29.703) | -20.40 (24.212)
  Change at 216 hours: number analyzed (Participants) | 4 | 3 | 6 | 2
  Change at 216 hours | -44.10 (35.056) | 13.87 (15.597) | -4.90 (43.425) | NA (NA) — Mean and SD were not determined because insufficient number of participants (<=2 participants) had data and therefore, summary statistics could not be performed, as was pre-specified in the analysis plan.
  Change at 288 hours: number analyzed (Participants) | 4 | 2 | 6 | 2
  Change at 288 hours | -38.40 (33.032) | NA (NA) — Mean and SD were not determined because insufficient number of participants (<=2 participants) had data and therefore, summary statistics could not be performed, as was pre-specified in the analysis plan. | 2.58 (32.591) | NA (NA) — Mean and SD were not determined because insufficient number of participants (<=2 participants) had data and therefore, summary statistics could not be performed, as was pre-specified in the analysis plan.
  Change at 648 hours: number analyzed (Participants) | 4 | 2 | 6 | 3
  Change at 648 hours | -34.30 (45.276) | NA (NA) — Mean and SD were not determined because insufficient number of participants (<=2 participants) had data and therefore, summary statistics could not be performed, as was pre-specified in the analysis plan. | 25.17 (30.641) | -26.93 (45.377)

15. Secondary Outcome: Change From Baseline in Von Willebrand Factor:Ristocetin Cofactor Activity (VWF:RCo) At Specified Timepoints
Description: Von Willebrand factor (vWF or VWF) is a protein that is one of several components of the coagulation system that work together, to stop bleeding within the body. VWF:RCo assay is a test that measures the activity of the VWF in a plasma sample in terms of how well it is able to clump platelets together in the presence of the antibiotic ristocetin. Change from baseline in vWF:RCo concentration was measured at different timepoints. Baseline was defined as the last non-missing measurement obtained prior to the date and time of the dose of IP. Change from baseline was calculated by subtracting the baseline value from the post-dose value.
Time Frame: Baseline (Pre-dose), 0.25, 1, 3, 8, 24, 72, 120, 168, 216, 288, and 648 hours post-dose
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Percentage of vWF RCo
Arm/Group | Placebo | TAK-755: 40 IU/kg | TAK-755: 80 IU/kg | TAK-755: 160 IU/kg
Number analyzed (Participants) | 4 | 3 | 6 | 4
Percentage of vWF RCo
  Change at 0.25 hours: number analyzed (Participants) | 4 | 3 | 5 | 4
  Change at 0.25 hours | -6.78 (8.107) | -7.40 (10.802) | -6.06 (14.134) | -3.50 (13.365)
  Change at 1 hour | -10.08 (11.346) | -7.80 (9.242) | 6.63 (31.637) | -4.60 (8.285)
  Change at 3 hours: number analyzed (Participants) | 4 | 3 | 5 | 3
  Change at 3 hours | -9.75 (5.047) | -20.80 (72.904) | -10.10 (7.833) | -7.00 (10.835)
  Change at 8 hours: number analyzed (Participants) | 4 | 3 | 5 | 3
  Change at 8 hours | 0.28 (34.209) | -34.80 (63.461) | -17.36 (34.424) | -8.00 (14.178)
  Change at 24 hours | 8.30 (5.582) | 20.07 (36.049) | 9.32 (18.590) | -1.20 (26.771)
  Change at 72 hours | -8.03 (8.176) | 20.17 (22.167) | 8.60 (9.908) | -11.30 (11.895)
  Change at 120 hours: number analyzed (Participants) | 3 | 2 | 6 | 4
  Change at 120 hours | 4.33 (15.284) | NA (NA) — Mean and SD were not determined because insufficient number of participants (<=2 participants) had data and therefore, summary statistics could not be performed, as was pre-specified in the analysis plan. | -32.33 (50.707) | -0.55 (11.301)
  Change at 168 hours: number analyzed (Participants) | 3 | 2 | 6 | 4
  Change at 168 hours | -9.87 (6.217) | NA (NA) — Mean and SD were not determined because insufficient number of participants (<=2 participants) had data and therefore, summary statistics could not be performed, as was pre-specified in the analysis plan. | 0.97 (7.227) | 15.00 (9.367)
  Change at 216 hours | -15.90 (20.132) | 13.20 (37.091) | 9.35 (8.005) | 7.08 (22.733)
  Change at 288 hours: number analyzed (Participants) | 4 | 2 | 6 | 4
  Change at 288 hours | -22.33 (11.712) | NA (NA) — Mean and SD were not determined because insufficient number of participants (<=2 participants) had data and therefore, summary statistics could not be performed, as was pre-specified in the analysis plan. | 8.58 (3.812) | 7.83 (36.533)
  Change at 648 hours: number analyzed (Participants) | 4 | 2 | 6 | 4
  Change at 648 hours | -17.03 (10.801) | NA (NA) — Mean and SD were not determined because insufficient number of participants (<=2 participants) had data and therefore, summary statistics could not be performed, as was pre-specified in the analysis plan. | 9.43 (10.112) | -12.83 (83.921)

16. Secondary Outcome: Change From Baseline in Platelet Count at Specified Timepoints
Description: Blood samples were collected to analyze platelet count. Baseline was defined as the last non-missing measurement obtained prior to the date and time of the dose of IP. Thechange from baseline was calculated by subtracting the baseline value from the post-dose value.
Time Frame: Baseline (Pre-dose), 3, 8, 24, 72, 120, 168, 216, 288, and 648 hours post-dose
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Placebo | TAK-755: 40 IU/kg | TAK-755: 80 IU/kg | TAK-755: 160 IU/kg
Number analyzed (Participants) | 5 | 4 | 6 | 4
10^9 cells per liter
  Change at 3 hours: number analyzed (Participants) | 5 | 4 | 5 | 4
  Change at 3 hours | -39.40 (35.795) | 3.50 (27.111) | -42.80 (27.151) | -32.00 (19.511)
  Change at 8 hours: number analyzed (Participants) | 5 | 4 | 5 | 3
  Change at 8 hours | -33.96 (29.535) | 11.40 (24.309) | -38.42 (33.679) | -23.77 (25.325)
  Change at 24 hours | -1.60 (38.946) | 22.88 (36.779) | -11.83 (55.654) | -18.50 (25.265)
  Change at 72 hours | -20.80 (61.378) | 36.35 (19.025) | -7.10 (81.770) | -40.75 (64.691)
  Change at 120 hours: number analyzed (Participants) | 4 | 3 | 5 | 4
  Change at 120 hours | 4.50 (100.018) | 40.83 (35.617) | 18.94 (104.933) | -47.25 (61.927)
  Change at 168 hours: number analyzed (Participants) | 5 | 3 | 6 | 3
  Change at 168 hours | -38.40 (94.648) | 22.33 (58.046) | 20.35 (122.803) | -73.33 (97.007)
  Change at 288 hours: number analyzed (Participants) | 4 | 3 | 6 | 4
  Change at 288 hours | -42.00 (97.060) | 17.67 (10.408) | 6.17 (105.447) | -50.75 (70.296)
  Change at 648 hours | -116.40 (232.119) | 29.00 (27.313) | 6.93 (77.027) | 3.75 (51.344)

17. Secondary Outcome: Change From Baseline in Plasma Free Hemoglobin at Specified Timepoints
Description: The plasma free hemoglobin test measures the level of hemoglobin in the plasma (that is, not contained within the red blood cells). Baseline was defined as the last non-missing measurement obtained prior to the date and time of the dose of IP. Change from baseline was calculated by subtracting the baseline value from the post-dose value.
Time Frame: Baseline (Pre-dose), 3, 8, 24, 72, 120, 168, 216, 288, and 648 hours post-dose
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Placebo | TAK-755: 40 IU/kg | TAK-755: 80 IU/kg | TAK-755: 160 IU/kg
Number analyzed (Participants) | 4 | 4 | 3 | 4
milligrams per deciliter (mg/dL)
  Change at 3 hours: number analyzed (Participants) | 4 | 4 | 2 | 4
  Change at 3 hours | -5.23 (21.732) | -8.98 (23.930) | NA (NA) — Mean and SD was not determined as the sample size (<= 2 observed values) were not sufficient to determine the Plasma Free Hemoglobin parameter. | -106.15 (216.380)
  Change at 8 hours: number analyzed (Participants) | 4 | 4 | 2 | 3
  Change at 8 hours | -11.28 (18.671) | -30.58 (34.219) | NA (NA) — Mean and SD was not determined as the sample size (<= 2 observed values) were not sufficient to determine the Plasma Free Hemoglobin parameter. | -147.80 (251.263)
  Change at 24 hours | -3.88 (21.390) | -34.28 (36.621) | -44.77 (47.417) | -105.95 (214.072)
  Change at 72 hours: number analyzed (Participants) | 4 | 3 | 3 | 4
  Change at 72 hours | -9.23 (22.105) | -44.93 (35.400) | -49.27 (47.550) | -108.30 (218.455)
  Change at 120 hours: number analyzed (Participants) | 3 | 2 | 3 | 4
  Change at 120 hours | -14.70 (27.120) | NA (NA) — Mean and SD was not determined as the sample size (<= 2 observed values) were not sufficient to determine the Plasma Free Hemoglobin parameter. | -47.47 (48.187) | -98.18 (226.371)
  Change at 168 hours: number analyzed (Participants) | 4 | 3 | 3 | 3
  Change at 168 hours | -10.60 (23.047) | -44.37 (50.024) | -41.37 (47.933) | -123.83 (274.097)
  Change at 288 hours: number analyzed (Participants) | 4 | 3 | 3 | 3
  Change at 288 hours | -8.05 (25.683) | -46.47 (43.714) | -46.67 (47.013) | 5.17 (4.319)
  Change at 648 hours: number analyzed (Participants) | 4 | 4 | 3 | 3
  Change at 648 hours | 13.30 (53.656) | -26.43 (45.465) | -43.83 (50.519) | -130.87 (265.316)

18. Secondary Outcome: Change From Baseline in Plasma Thrombospondin Levels at Specified Timepoints
Description: Change from baseline in plasma thrombospondin levels over time was reported. Baseline was defined as the last non-missing measurement obtained prior to the date and time of the dose of IP. Change from baseline was calculated by subtracting the baseline value from the post-dose value.
Time Frame: Baseline (Pre-dose), 3, 8, 24, 72, 120, 168, 288, and 648 hours post-dose
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Groups:
- Placebo; TAK-755: 160 IU/kg: Participants with SCD at their baseline health received a single IV infusion of TAK-755 at a dose level of 160 IU/kg on Day 1 and followed for up to 28 days.
Arm/Group | Placebo | TAK-755: 40 IU/kg | TAK-755: 80 IU/kg | TAK-755: 160 IU/kg
Number analyzed (Participants) | 5 | 4 | 6 | 4
nanograms per milliliter (ng/mL)
  Change at 3 hours: number analyzed (Participants) | 5 | 4 | 5 | 4
  Change at 3 hours | 840.4 (3979.24) | -628.5 (1420.49) | -1177.2 (1730.05) | -736.3 (860.29)
  Change at 8 hours: number analyzed (Participants) | 5 | 4 | 5 | 3
  Change at 8 hours | -1892.8 (3500.43) | -604.5 (1763.64) | -1471.8 (1274.07) | -1290.0 (1060.98)
  Change at 24 hours | -934.0 (1815.42) | -408.0 (1140.98) | -1077.0 (1699.60) | -1567.8 (957.61)
  Change at 72 hours | -701.4 (2560.18) | -651.8 (1208.59) | -1080.0 (1945.58) | -1406.0 (843.31)
  Change at 120 hours: number analyzed (Participants) | 4 | 3 | 6 | 4
  Change at 120 hours | -1075.0 (1357.88) | -1428.7 (1892.45) | -331.8 (3735.24) | 1351.8 (5880.93)
  Change at 168 hours: number analyzed (Participants) | 4 | 3 | 6 | 4
  Change at 168 hours | -3886.0 (3999.22) | -847.0 (1728.41) | -1623.7 (1569.60) | -687.5 (1373.36)
  Change at 288 hours: number analyzed (Participants) | 4 | 3 | 6 | 4
  Change at 288 hours | -103.0 (1974.37) | -482.0 (1150.09) | -1290.7 (1723.60) | -903.5 (1232.02)
  Change at 648 hours | -2857.0 (4236.96) | -766.0 (1948.34) | -909.7 (1082.66) | 525.5 (3358.11)

ADVERSE EVENTS:
Time Frame: From date of signing informed consent up to end of study visit (Day 28)
Description: SAS included all participants randomized and who received any dose of IP.
Groups:
- Placebo: Participants with SCD at their baseline health received a single IV infusion of placebo matched to TAK-755 at 3 dose levels of 40 IU/kg, 80 IU/kg, and 160 IU/kg on Day 1 and followed up for to 28 days.
Arm/Group | Placebo | TAK-755: 40 IU/kg | TAK-755: 80 IU/kg | TAK-755: 160 IU/kg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/4 | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 2/5 | 2/4 | 4/6 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=5) | TAK-755: 40 IU/kg (N=4) | TAK-755: 80 IU/kg (N=6) | TAK-755: 160 IU/kg (N=4)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=5) | TAK-755: 40 IU/kg (N=4) | TAK-755: 80 IU/kg (N=6) | TAK-755: 160 IU/kg (N=4)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2021-07-12): https://cdn.clinicaltrials.gov/large-docs/60/NCT03997760/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-04): https://cdn.clinicaltrials.gov/large-docs/60/NCT03997760/SAP_001.pdf